CLINICAL TRIAL: NCT00802581
Title: Does Ensuring Circumferential Local Anesthetic Spread Improve the Success of Ultrasound Guided Sciatic Nerve Block at the Popliteal Fossa?
Brief Title: Circumferential Spread of Anesthetic and Success in Sciatic Nerve Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-0728-B
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2010-05

CONDITIONS: Sciatic Nerve Blockade for Foot/Ankle Surgery
Keywords: sciatic nerve block; local anesthetic; lidocaine; ankle surgery; foot surgery; ultrasound-guided regional anesthesia; circumferential spread; anesthetic infiltration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ensuring circumferential spread of local anesthetic around the sciatic nerve.
  Interventions: Procedure: Circumferential spread of local anesthetic
- 2 (Active Comparator): Single shot injection of local anesthetic near the sciatic nerve will be performed, without ensuring circumferential spread.
  Interventions: Procedure: Non-circumferential spread of local anesthetic

INTERVENTIONS:
Procedure: Circumferential spread of local anesthetic — The anesthetist will ensure, under ultrasound guidance, that local anesthetic (1 mL of 1% lidocaine) surrounds the sciatic nerve.
  Arms: 1
Procedure: Non-circumferential spread of local anesthetic — The anesthetist will perform a "single shot" injection of local anesthetic (1 mL of 1% lidocaine) near the sciatic nerve under ultrasound guidance, without ensuring circumferential spread around the nerve.
  Arms: 2

SUMMARY:
Current practices when performing any peripheral nerve block may or may not involve ensuring circumferential spread of local anesthetic around the nerve. Ensuring circumferential spread can involve several redirections of the needle above and below the nerve, and potentially could result in either more discomfort for the patient or an increased chance of inadvertent direct trauma to the nerve. Not ensuring spread around the nerve may result in a slower and less complete blockade. The investigators suspect that by ensuring complete spread around the nerve, the speed of block onset would be quicker because it avoids the loss due to diffusion time.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking
2. ASA physical status I-III
3. 18-85 years of age, inclusive
4. 50-110 kg, inclusive
5. 150 cm of height or grater
6. Scheduled for elective foot or ankle surgery

Exclusion Criteria:

1. Contraindications to sciatic nerve block (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the popliteal area)
2. Significant peripheral neuropathy or neurologic disorder affecting the lower extremity
3. Pregnancy
4. Contraindications to, allergies to, and/or past adverse reactions to study medications (local anesthetics, opioid analgesics)
5. History of alcohol or drug dependency/abuse
6. History of long term opioid intake
7. History of significant psychiatric conditions that may affect patient assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Onset time of sciatic nerve blockade. | Every 5 minutes for 30 minutes after anesthetic injection

SECONDARY OUTCOMES:
Block success, time required to perform block, complications/adverse events, number of needle passes, patient discomfort | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada